Title of Study: Toileting at Night in Older Adults: Light to Maximize Balance, Minimize Insomnia

NCT number: NCT01350505

Date of document: 9/26/18

## Initial analysis plan

To test our Primary Hypothesis that a long wavelength light stimulus delivered at night will improve gait and not change alertness, we will examine stride-to-stride variability in speed and change in EEG delta power as our two primary outcome measures. Statistical significance will be determined with independent repeated measure analyses of variance (ANOVA) with *post hoc t*-tests. Our *a priori* hypothesis is that gait will be progressively improved such that dim light < orange light = room light and that alertness will be improved such that dim light = orange light < room light.